CLINICAL TRIAL: NCT05319808
Title: Rehabilitation for Whiplash Associated Disorders; a Randomized Clinical Trial
Brief Title: Rehabilitation for Whiplash Associated Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Iceland (Other)
Collaborators: Empowered Health (Unknown); Reykjavik University (Other); Landspitali University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UI-123218
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Whiplash Injury of Cervical Spine
Keywords: Whiplash-Associated Disorders; Car-collision; Kinaesthesia; Telehealth; Motor Control; Treatment; Exercises; Manual Therapy; Objective measurements
MeSH Terms: conditions — Motor Activity | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Two groups will receive physiotherapy. Both will receive a "hands-on" individualized treatment of manual therapy. The "hands-off" treatment differs between groups and goes as follows:
  Group A will receive a novel, remote computer based cervical joint positioning exercise and cervical kinaesthesia exercise program with a 6-month follow-up.
  Group B will receive a non-computer based exercise regime at the need of each individual (pragmatic approach). This group will not be followed up on their exercises post intervention but will be encouraged to continue doing their exercises. They will be asked during follow-up measurements if they have been doing their exercises.
  The "treatment as usual" group (group C) will/will not receive treatment at his/her own choice and/or convenience and without any instructions from research staff to reflect general practice. In addition to follow-up assessments, data will be collected which asks about treatment modalities used.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Telehealth using NeckCare equipment
  Interventions: Other: Manual therapy; Device: Telehealth exercises
- Group B (Active Comparator): Exercises without telehealth intervention
  Interventions: Other: Manual therapy; Other: Non-computer based exercises
- Group C (No Intervention): No intervention provided by the researchers

INTERVENTIONS:
Other: Manual therapy — Individualized treatment of manual therapy provided by MT PTs, graduates from Curtin University of Technology, Perth, Australia (2008)
  Arms: Group A; Group B
Device: Telehealth exercises — A novel, remote computer based cervical joint positioning exercise and cervical kinaesthetic exercise (CKE) program. A technical consultant monitors the data from the remote exercises and inform the PTs if someone has not done their exercises in over 2 weeks during the study period so subjects can be encouraged with a friendly reminder.
  Arms: Group A
Other: Non-computer based exercises — Home-exercises in the need of each subject (pragmatic approach) taught by MT PTs, graduates from Curtin University of Technology, Perth, Australia (2008)
  Arms: Group B

SUMMARY:
Individuals (n=180) with subacute (<1 month, >3 months) WAD grade I and II with medium to high-risk symptoms of working age will be randomized into three groups with block randomization in a prospective, assessor-blinded randomized controlled trial. Two primary intervention groups (A and B) will receive manual therapy (MT) in the same out-patient clinic. In addition, group A will receive a remote, novel, computer-based cervical kinaesthetic exercise program starting at visit two, whereby quality and quantity of exercise performance, as well as compliance (frequency and duration), will be registered into the physical therapy clinic's system for evaluation. Group B will receive neck exercises (not computer-based) provided by the corresponding physical therapist. Group A will continue remote exercise therapy until 6 months post baseline measurements regardless of whether they are still being treated in-clinic or discharged.

Hypothesis 1.a.: Internet-based neck-specific CKE combined with in-clinic manual therapy and exercises will be superior to manual therapy and exercises alone at a physiotherapy clinic (i.e., treatment A is superior to treatment B) for self-reported and measured (movement performance) outcome measures.

Hypothesis 1.b.: Improvements in self-reported outcomes will positively correlate with outcomes of movement performance testing, as will the pre- to post-intervention changes from baseline to follow-up assessments.

The groups will be compared to a "treatment as usual" group (C). Objective measures include measurements for motor control, proprioception, and cervical range of motion. Neck disability and pain intensity, general health, self-perceived handicap, and physical, emotional and functional difficulties due to dizziness will be measured using questionnaires. Short-term effects will be measured at 10-12 weeks and long-term effects at 6- and 12-months post baseline measurements.

Hypothesis 2.a.: Participants of groups A and B will improve significantly more than those in group C for subjective and objective outcome measures.

DETAILED DESCRIPTION:
QUALITY ASSURANCE PLAN:

PhD student will monitor the data and guarantee high data quality. Data will be protected according to the Act on Data Protection and the Processing of Personal data (Icelandic law) and stored at the University Hospital or at a secure NeckCare database. Data will be registered into Microsoft Excel and shared through a secure network with other researchers to promote transparency.

DATA CHECKS:

Data will be checked for outliers.

SOURCE DATA VERIFICATION:

N/A

DATA DICTIONARY:

WAD: whiplash-associated disorders; MVC: motor vehicle collision; VR: virtual reality; NDI: neck disability index; ROM: range of motion; PTs: physiotherapists; MT: manual therapy; CKE: cervical kinaesthetic exercise; IT: information technology; IoT: internet of things; IMU: inertial monitoring unit; VAS: visual analog scale; SF-36: short form 36 item health survey; DHI: dizziness handicap inventory; CSI: central sensitisation inventory; CS: central sensitization; ToT: time on target; CI: confidence interval; MCIC: minimal clinically important changes.

STANDARD OPERATION PROCEDURES:

A total of 180 subjects (60 from each of the three groups) will be recruited through the databases of The Emergency Department of Landspitali University Hospital, Reykjavik, Iceland via phone call.

Subjective and objective outcome measures will be collected by a PhD student. In addition to questionnaire and clinical outcome measures, the pharmaceutical database of the Directorate of Health in Iceland will be accessed for data on subjects' drug use.

Data will be analysed by the PhD student using Microsoft Excel and R, a free software environment for statistical computing and graphics.

The PhD student will be responsible for reporting adverse events and change management.

SAMPLE SIZE ASSESSMENT:

Sample size and power regarding group differences will be calculated based on the primary outcome NDI. To detect a clinically relevant improvement of 8% in the NDI, 40 participants are needed in each group for 80% power. For non-inferiority tests, the significance level will be set to 5% (p > 0.05) which corresponds to the one-sided confidence interval (95% CI). To ensure that enough people are in each group after dropouts, for prediction analyses and the opportunity for subgroup analyses, 60 participants will be included in each group (n=180).

PLAN FOR MISSING DATA:

If data will be found to be missing by any reason, each incident will be assessed by the PhD student and her advisors. Imputation methods may be used, the subject involved may be asked to come back in for a measurement or answer questionnaires again (depending on the time that has passed from the measurement/questionnaires until data is discovered missing) or the subject involved will be removed from the study.

STATISTICAL ANALYSIS PLAN:

Data analyses and statistics Database monitoring will be performed by the primary researcher and statisticians involved, independent of sponsors and competing interests. Background data will be assessed after all subjects have completed their baseline measurements.

Background data and association of self-reported and clinical measures Background data will be evaluated with descriptive statistics and differences in baseline data determined using t-tests and (M)ANOVA (mean and standard deviation) or non-parametric tests where appropriate. Association of self-reported measurements and clinical measures will be assessed for baseline, 10-12-week, 6-month and 12-month measurements using Pearson or Spearman correlation depending on the distribution of the data. Subgroup analyses of CPS may possibly be performed.

Effectiveness of therapy Analyses will be performed primarily on an intention-to-treat basis (as individuals being randomized into the groups) and secondarily on a per protocol basis (individuals who fulfilled the programme for at least 50%). Imputation methods may be used when deemed to have additional value. Linear mixed models with time as a repeated factor will be used to assess the effect of treatment for each outcome. Correlation over time, within the PT and prognostic factors will be accounted for. Estimates of the effect of the intervention will be obtained by constructing linear contrasts to compare the mean change in outcome for each measurement (subjective and objective) to each time point between treatment groups and between each treatment group compared to control group. The main dependent variable will be score on NDI with independent fixed factors time (baseline, 10-12-week, 6-month, and 12-month) and group (A, B and C). If the non-inferiority of C to A or of C to B is concluded based on the 95% CI, a test of the superiority of C to A or of C to B will be performed as suggested by Lesaffre (see reference list). The variation in response to intervention (heterogeneity of treatment effect) will be evaluated using regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* subacute (>1 month, <3 months) neck problems corresponding to WAD grades I-II verified by WhipPredict
* medium to high risk symptoms (NDI score >32% OR subject is >36 years old) OR VAS score >4/10
* within daily reach of a computer/tablet/smartphone and Internet
* showed neck symptoms within the first week following the car collision (i.e. neck pain, neck stiffness)

Exclusion Criteria:

* WAD grades III-IV
* considerable degree of known or suspected physical pathology (Myelopathy, Spinal tumours, Spinal infection, Ongoing malignancy, Cervical spine surgery, Severe neck problems within their medical history which resulted in sick leave for more than a month in the year before the current whiplash injury, Other illness/injury that may prevent full participation from being feasible, Lack of ability to either understand or write Icelandic, Severe obesity (body mass index; BMI > 35), Pregnancy)
* unable to complete the assessment

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Neck disability index (NDI) | 5 minutes
  the NDI is a 10-item self-report questionnaire that has been shown to demonstrate good validity and reliability. Each section is scored on a 0 to 5 rating scale, higher score represents more neck pain related disability.
Visual Analog Scale (VAS) | 1 minutes
  Neck pain intensity during the past week prior to each measurement measured by a 100 mm visual analogue scale (VAS) with 0mm representing "no pain" and 100mm representing "worst pain imaginable
Butterfly Test | 5 minutes
  * Procedure: The subject tracks an unpredictable path as accurately as possible using head movement to manipulate the on-screen cursor. There are different trajectories with increasing difficulty. The subject repeats each trajectory path 3 times.
  * Metrics: (1) Amplitude Accuracy (AA): the absolute distance (radius) in mm between the cursor that represents the head position and the target. (2) Time On Target (ToT): the percentage of time the cursor that represents the head position spends in a mathematically determined, invisible free zone around the target. (3) Smoothness of Movement Index (SMI): The index is calculated based on the third positional derivative with respect to time and is scaled between 0 and 5 with 0 being the best and 5 being the worst.
Whole Cervical Range of Motion (ROM) Test | 5 minutes
  * Procedure: The subject turns their head using four different types of movements: flexion, extension, rotation (left/right) and lateral flexion (left/right) to measure the maximum range ROM. Each movement is repeated 3 times.
  * Metrics: An average degree value and standard deviation of the 3 measurements for each movement type.
Head Neck Relocation Test (HNRT) | 5 minutes
  * Procedure: While blindfolded, the subject is asked to find their "neutral" position. The subject then turns their head to rotate left/right and up/down and attempts to return to the neutral/initial position following each movement, the subject informs the researcher by saying a simple "ok" when he believes he has reached the neutral position. The researcher marks this with one mouse click.
  * Metrics: (1) Accuracy Error measures the deviation in degrees from the initial position; (2) Constant Error measures under-/overshooting; and (3) Variable Error measures the precision of the head posture.

SECONDARY OUTCOMES:
SF-36 Health Survey (SF-36) RAND version | 10 minutes
  SF-36 is the most frequently recommended questionnaire to rate general mental health for patients with chronic musculoskeletal disorders. It's a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting, and the 36 items tap eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0 to 100 range where higher score defines a more favorable health state.
Dizziness Handicap Inventory (DHI) | 5 minutes
  the DHI is a 25-item self-assessment inventory designed to evaluate the self-perceived handicapping effects imposed by dizziness. Each item is scored on a 0 to 4 rating scale, with higher score representing more self-perceived handicapping.
Central Sensitization Inventory (CSI) | 5 minutes
  the CSI is a self-reported tool to assess symptoms of CS (central sensitization). The list includes 25 items about CS-related symptoms, scored on a five-point Likert scale from 0-4. Higher total scores reflect higher CS symptomology

OTHER OUTCOMES:
Background data, questionnaire | 7 minutes
  Background data that will be collected will include age, sex, date of birth, information on when the accident occurred and how, first symptoms, former healthcare, education, occupational classification, income, and information on insurance claim status. Furthermore, during the 6-month and 12-month follow-up participants will also be asked to give information on if they have met with a health care practitioner for treatment other than those of this study

CONTACTS AND LOCATIONS:
Overall Officials: Kristín Briem, PhD, Study Chair — University of Iceland
Locations (4):
- Iceland (4):
  - K!M Rehabilitaion, Kopavogur
  - University of Iceland, Reykjavik
  - Landspítali University Hospital, Reykjavik
  - Hæfi Physiotherapy, Reykjavik

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lesaffre E. Superiority, equivalence, and non-inferiority trials. Bull NYU Hosp Jt Dis. 2008;66(2):150-4. PMID 18537788
- [Derived] Ragnarsdottir H, Briem K, Oddsdottir GL. Effects of a Novel Web-Based Sensorimotor Exercise Program for Patients With Subacute Whiplash-Associated Disorders: Protocol for a Randomized Clinical Trial. Phys Ther. 2023 Aug 1;103(8):pzad063. doi: 10.1093/ptj/pzad063. PMID 37338163